CLINICAL TRIAL: NCT05505435
Title: Continuation Rates of Self-administered Subcutaneous Depot Medroxyprogesterone Acetate and Provider-administered Intramuscular Depot Medroxyprogesterone Acetate in Patients Seeking Post-abortion Contraception
Brief Title: Continuation of Subcutaneous and Intramuscular Depot Medroxyprogesterone Acetate in Post-abortion Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Ashley Turner, MD, Assistant Professor, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00216775
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Contraception
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DMPA-SC (Active Comparator): self-administered subcutaneous depot medroxyprogesterone acetate 104 mg
  Interventions: Drug: Depot-Medroxyprogestereone Acetate
- DMPA-IM (Active Comparator): provider-administered intramuscular depot medroxyprogesterone acetate 150 mg
  Interventions: Drug: Depot-Medroxyprogestereone Acetate

INTERVENTIONS:
Drug: Depot-Medroxyprogestereone Acetate — subcutaneous depot medroxyprogesterone acetate
  Arms: DMPA-SC
Drug: Depot-Medroxyprogestereone Acetate — intramuscular depot medroxyprogesterone acetate
  Arms: DMPA-IM

SUMMARY:
Multiple prior studies have compared self-administered Subcutaneous Depot Medroxyprogesterone Acetate(DMPA-SC) to both provider-administered DMPA-SC and Intramuscular Depot Medroxyprogesterone Acetate (DMPA-IM) and found that continuation rates for self-administered DMPA-SC are higher. Thus far, studies investigating self-administered DMPA-SC have focused on patients presenting for contraception. Self-administered DMPA-SC has not been widely studied in patients seeking abortion and has been more extensively studied in international settings than in the US. The project will be a prospective cohort study of patients at a large, free-standing abortion clinic in Chicago, Illinois. Patients who indicate that they desire DMPA for post-abortion contraception will be recruited. They will choose either provider-administered DMPA-IM or self-administered DMPA-SC. Patients in both groups will complete a baseline survey that will collect demographic and clinical characteristics. Patients who choose self-administered DMPA-SC will receive self-injection teaching from study staff and will self-inject their first dose of DMPA-SC in the clinic. Patients who choose provider-administered DMPA-IM will receive their first dose of DMPA-IM in the clinic. Both groups will receive a prescription for three additional doses of DMPA and will receive an injection calendar. Study participants will receive a reminder prior to the start of the injection window for their second and third doses. After the injection window for the second and third doses closes, participants will complete follow up surveys. These surveys will assess whether patients received the subsequent doses of DMPA, reasons for discontinuing DMPA for patients who did not receive a dose, pregnancy status, and patient satisfaction with DMPA use. Follow up will be primarily via secure text messaging application with phone calls, email, and mail reserved for patients who cannot or prefer not to be contacted via text message. The primary outcome is continuation rates of DMPA-IM and DMPA-SC at 3 and 6 months after initiation. Secondary outcome measures include pregnancy, adverse effects, and patient satisfaction. We will also determine associations between patients' demographic and clinical characteristics and continuation of DMPA. This project will generate evidence that will support expanding access to DMPA-SC and providing patient education on self-injection, allowing for increased patient contraceptive autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient planning DMPA for post-abortion contraception.

Exclusion Criteria:

* Patient cannot speak and read English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
DMPA continuation rate | 6 months
  Participant use of DMPA 6 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Family Planning Associates, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No